CLINICAL TRIAL: NCT04777149
Title: Random Noise Stimulation to Enhance Corticomotor Drive for Improved Hand Function
Brief Title: Random Noise Stimulation to Enhance Cortical Drive & Improve Hand Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 762
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injuries; Tetraplegia; Cervical Spinal Cord Injury
Keywords: Non-invasive brain stimulation; Hand function; Random noise
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Wash-in control design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcranial Random Noise Stimulation (tRNS) (Experimental): Participants in this group will receive a combined intervention (3 days of tRNS during functional task practice and 3 days of sham-stimulation during functional task practice).
  Interventions: Other: transcranial Random Noise Stimulation (tRNS); Other: sham-stimulation
- transcranial Direct Current Stimulation (tDCS) (Active Comparator): Participants in this group will receive a combined intervention (3 days of tDCS during functional task practice and 3 days of sham-stimulation during functional task practice).
  Interventions: Other: transcranial Direct Current Stimulation (tDCS); Other: sham-stimulation

INTERVENTIONS:
Other: transcranial Random Noise Stimulation (tRNS) — Two electrodes will be placed over the targeted areas on participant's head. A current of random frequency and intensity will be delivered. TRNS will be applied during the first 20 min of functional task practice.
  Arms: transcranial Random Noise Stimulation (tRNS)
Other: transcranial Direct Current Stimulation (tDCS) — Two electrodes will be placed over the targeted areas on participant's head. A continuous low intensity current will be delivered. TDCS will be applied during the first 20 min of functional task practice.
  Arms: transcranial Direct Current Stimulation (tDCS)
Other: sham-stimulation — Two electrodes will be placed over the targeted areas on participant's head. A continuous low intensity current will be delivered for 1- 2 min.

SUMMARY:
Cervical spinal cord injury (SCI) results in hand and arm function impairments and decreased independence in performance of daily activities such as bathing, eating, dressing, writing, or typing. Recent approaches that involve the application of non-invasive brain stimulation have the potential to strengthen the remaining connections between the brain and the spinal cord for improved hand function. Combining brain stimulation with performing upper limb functional tasks may further increase the ability of individuals with tetraplegia to use their hands. The purpose of this study is to investigate if "random noise", a special type of brain stimulation that most people cannot feel, can be used to enhance upper limb function in individuals with spinal cord injury. Specifically, the investigators will examine if a combined treatment protocol of random noise and fine motor training results in greater improvements in motor and sensory hand function compared to fine motor training alone.

DETAILED DESCRIPTION:
Cervical spinal cord injury (SCI) results in upper extremity (UE) functional impairments that can restrict independence, social participation, and overall quality of life. Evidence shows that short duration of non-invasive brain stimulation (NIBS) can strengthen the transmission of information through the spared corticospinal pathways and improve UE functional recovery in individuals with tetraplegia. Transcranial direct current stimulation (tDCS), which is a clinically accessible NIBS approach, has been used to modulate cortical plasticity and improve hand function. However, the high variability in the reported effects of tDCS raises questions about its clinical value and highlights the need to investigate more robust NIBS protocols. Transcranial random noise stimulation (tRNS) is a novel NIBS approach that produces more consistent facilitatory effects compared to tDCS. TRNS delivers a low alternating current with a continuously changing intensity over a wide frequency range. Further, tRNS has excellent tolerability and no risk of skin burns since it is a polarity independent stimulation approach. When tRNS is applied over the motor cortex, it increases cortical excitability in the hand representation area and enhances motor learning in healthy adults. Despite the potential promise of tRNS in increasing corticomotor drive for improved motor performance, its application in persons with SCI is novel. Therefore, in this study, the investigators propose to use tRNS to augment the therapeutic effects of functional task practice (FTP). Our aim is to compare the efficacy of a 3-day tRNS+FTP protocol on cortical excitability, UE motor, and sensory function to tDCS+FTP and to sham-stimulation+FTP in individuals with tetraplegia.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury level above C8
* ASIA Impairment Scale (AIS) classification level: C, D
* Time since injury: ≥ 1 year
* Active intrinsic hand muscles in at least one UE
* Active extrinsic hand muscles in both UE
* Ability to follow multiple step commands
* Ability to communicate pain or discomfort
* Willingness to participate in testing
* Ability to obtain informed consent

Exclusion Criteria:

* Implanted metallic device in the head and/ or pacemaker
* History of seizures
* History of severe headaches
* Severe contractures of UE that would limit participation in FTP
* Prior tendon or nerve transfer surgery
* Received Botulinum toxin injection in the tested UE in the last 3 months
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Change in Cortical excitability | Baseline; Post Testing Week 1; Post Testing Week 2
  The communication between brain and spinal cord will be evaluated. Sensors that detect muscle activity will be placed over hand muscles. Pulses of stimulation will be applied to the head using a type of non-invasive brain stimulation called transcranial magnetic stimulation (TMS). The size of the muscle response will be recorded.
Change in Strength (key pinch and grasp strength) | Baseline; Post Testing Week 1; Post Testing Week 2
  Key pinch and grasp strength will be assessed using a dynamometer.
Change in Sensory function (sensation subtest of the Graded Redefined Assessment of Strength Sensibility and Prehension) | Baseline; Post Testing Week 1; Post Testing Week 2
  Semmes and Weinstein Monofilaments will be applied on 3 dorsal and palmar sensory test locations in each hand. Each location is scored from 0 to 4.

SECONDARY OUTCOMES:
Change in Unimanual function (Grasp and Release Test) | Baseline; Post Testing Week 1; Post Testing Week 2
  Participants will be required to grasp, move, and release six objects of different size and weight. For each task, the number of successful and unsuccessful attempts is 30s will be recorded.
Change in Bimanual function (Chedoke Arm and Hand Activity Inventory) | Baseline; Post Testing Week 1; Post Testing Week 2
  This test consists of 9 functional tasks that require bimanual coordination. Each item is graded on a 7-point activity scale with higher scores suggesting better bimanual function.
Change in Sensory Function (revised Nottingham Sensory Assessment) | Baseline; Post Testing Week 1; Post Testing Week 2
  Tactile sensation, proprioception, stereognosis, and two-point discrimination will be tested. Higher scores indicate better sensory function.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Zarkou, PT,MS,PhD, Principal Investigator — Shepherd Center, Atlanta GA
Locations (1):
- Shepherd Center, Atlanta, Georgia, United States